CLINICAL TRIAL: NCT01131663
Title: Design and Development of an Infant's Oriented Face Mask
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Israel Amirav, Ziv Medical Center
Other Study IDs: 0063-09-ZIV
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Infant
Keywords: Infants, aerosol, acceptance, face mask, drug delivery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Face masks are used for many respiratory care applications such as anaesthesia, resuscitation, and aerosol therapy. None of the currently available face mask for infants and young children are specifically designed and developed for infants. The aim of this study is to design, develop and test the first infant's oriented face mask.

To achieve this ultimate goal we will first define appropriate sizes of infants' faces that would be used as templates for the design and development of optimally fitted model masks. In the next stage we will use these masks and incorporate the infants' own soother (pacifier) into a new SootherMask (SM). In the last part of the study we will compare acceptance levels between Soothermask (SM) and a conventional commodity masks without a pacifier.

DETAILED DESCRIPTION:
Not all face masks are "born equal" and care must be taken in mask design, particularly for the early pediatric age group. Unfortunately, facemasks provided for infants and young children have been merely smaller versions of those used for adults with little consideration given to their special needs

We believe that a major advance in answering the needs of infants rely in making the mask more friendly user by making sucking on the infant's soother an integral part of the newly developed mask. This is based on the following premises:

1. Sucking is a vital feeding and soothing activity of infants. Incorporating sucking into the act of aerosol delivery greatly reduces the fear engendered and inconvenience of putting an obtrusive mask on the infant's face.
2. Linking the mask to the sucking action ensures a tight seal between the mask and the face. Every time the baby sucks on the pacifier or the bottle nipple, the mask is pressed onto the face by atmospheric pressure thus ensuring a good mask to face seal. This then also ensures that the aerosol that has been sprayed into the holding chamber will be drawn into the baby's lungs through the nose with each inspiration.
3. The material of the mask's rim is relatively wide, soft, corrugated and is thus highly flexible. This makes the mask easily compressible without overdue force on the infant's face. Thus, the act of sucking attracts the mask to the child's face, assists in achieving a good seal and compresses it thus substantially reducing the dead space volume of the mask.

The ultimate goal of the present study is to answer these specific needs of infants and to develop an appropriate infant's oriented face mask. In order to achieve this goal the study will have three specific objectives.

Objective #1 Define morphometric data of infants' faces Objective #2 Design and develop an optimally adapted face mask SootherMask (SM) based on the morphometric results Objective #3 Compare the acceptance levels between Soothermask (SM) and a conventional commonly used masks without a pacifier.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent

Exclusion Criteria:

Non cooperation with procedure

Max Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: hospitals,primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Acceptance levels of new infant face mask | 10 minutes
  Infants will be offered two sets of simulated treatment options at random order:
  Placebo treatment by nebulizer (half the group) or by Valved Holding Chamber (VHC) (the other half) through the SM followed by placebo treatment by nebulizer (half the group) or by VHC (the other half) through the conventional mask.
  Treatments will be done sequentially at random order while the procedure is being captured and recorded on video. The video clips will be analyzed later off site and will be coded according to the scale in the scoring form to compare between acceptance levels of the two face masks.

CONTACTS AND LOCATIONS:
Overall Officials: Israel Amirav, MD, Principal Investigator — Ziv Medical Center
Locations (2):
- Israel (2):
  - Ziv Medical center, Safed
  - Pediatric Department, Ziv Medical Center, Safed